CLINICAL TRIAL: NCT04990739
Title: A Phase 1 Open Label, Multicenter Study of MTB-9655, an Inhibitor of ACSS2, in Patients With Advanced Solid Tumors
Brief Title: Study of MTB-9655, an Inhibitor of ACSS2, in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MetaboMed Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTB-9655-101
Record Dates: First submitted 2021-07-08; First posted 2021-08-04 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumor
Keywords: metastatic; ACSS2 inhibitor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Initial dose escalation will use an accelerated titration scheme followed by a 3+3 dose escalation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Part A Dose-Escalation and Part B RP2D Dose-Expansion (Experimental): Study has two parts:
  1. Part A Dose-Escalation will evaluate MTB-9655 monotherapy administered in 21 days cycle,and will be conducted in 2 stages (accelerated titration and dose-escalation).
     The first stage will consist of accelerated titration in single-patient cohorts for the initial two dose levels.
     In the second stage, a conventional 3+3 schema using a modified Fibonacci dose titration strategy will be implemented. The first dose at every dose level and in every patient will be administered under close medical supervision, and the patients will be hospitalized for approximately 24 hours.
     Up to 30 participants will participate in this dose escalation arm.
  2. Part B dose-expansion will further explore the safety, PK and preliminary efficacy of MTB-9655 at the RP2D. The RP2D level will be no higher than the MTD identified in Part A.
  Interventions: Drug: MTB-9655

INTERVENTIONS:
Drug: MTB-9655 — MTB-9655 is an orally available investigational product that is highly potent as it exhibits selectivity as an ACSS2 inhibitor when tested against a panel of related enzymes. MTB-9655 is formulated as a powder blend in a hydroxypropyl methylcellulose (HPMC) capsule and is presented as 25 mg and 100 mg strengths for oral administration.
  Patients will receive MTB-9655, by mouth daily in 21-day treatment cycles,either 1 hour before mealtime or 2 hours after mealtime.

SUMMARY:
MetaboMed is developing MTB-9655, an orally bioavailable, first-in-class small molecule inhibitor of the human Acetyl coenzyme A (Acyl-CoA) synthetase short chain family member 2 (ACSS2) enzyme, as a potential treatment for patients with cancer.

This study is a Phase 1,First-in-Human (FIH), open-label dose-escalation study of MTB-9655 given daily as a single oral (PO) agent. Up to 30 patients with locally advanced, unresectable and/or metastatic solid tumor(s) are expected to be enrolled in the dose-escalation portion (Part A). The study will be conducted at 1 to 2 sites in the United States and Israel.

DETAILED DESCRIPTION:
This Phase 1 First-in-Human (FIH) study is to initiate clinical development of MTB-9655 in patients with advanced solid tumors who have failed or refused standard treatment, or who have a tumor for which no therapy of proven efficacy exists. This study of MTB-9655 may consist of 2 parts: a dose-escalation part to establish a safe and tolerable dose of MTB-9655 in patients with advanced or metastatic solid tumors for which no standard therapy is available or standard therapy has failed (Part A), and a dose expansion phase (Part B) which may be initiated at the Sponsor's discretion after the maximum tolerated dose (MTD) (or recommended Phase 2 dose [RP2D]) has been determined in the dose-escalation (Part A), and with approval of an amendment to the protocol. This study will be the basis for future studies. The study will identify the safety and tolerability of MTB-9655 when administered on a continuous dosing schedule (given by mouth on a 21-day schedule).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Patient is at least 18 years-of-age at the time of signature of the informed consent form (ICF).
3. Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
4. Patient must have a confirmed diagnosis of locally advanced, unresectable and/or metastatic solid tumor(s), have failed standard treatment, or refuse standard treatment, or have a tumor for which no therapy of proven efficacy exists, or a tumor that is not amenable to standard therapies.
5. Patient has measurable disease on imaging based or non-measurable disease.
6. Patient will be requested to provide a fresh pre-treatment biopsy specimen, otherwise they are required to provide an archival diagnostic tumor sample that is <1 year old.
7. Patient has a life expectancy ≥3 months according to the Investigator's judgment.
8. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test at screening within 72 hours of first dose of MTB-9655. In addition, WOCBP are required to use two forms of acceptable contraception.
9. Male patients with WOCBP partners must agree to use highly effective contraceptive measures throughout the study starting with screening visit through 120 days after the last dose.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Treatment with any of the following:

   * Any systemic anti-cancer chemotherapy, small molecule, biologic, or hormonal agent from a previous treatment regimen or clinical study within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. At least 10 days must have elapsed between the last dose of such agent and the first dose of study drug.
   * Wide-field radiotherapy administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug.
   * Major surgery(excluding placement of vascular access) within 3 weeks of first dose of study drug.
   * Prior treatment with other drug with the same mechanism of action (directed to ACSS2).
   * Receiving systemic corticosteroid therapy 1 week prior to the first dose of study drug or receiving any other form of systemic immunosuppressive medication for medically significant acute or chronic conditions.
2. Persistent toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade >1 severity that is related to prior therapy.
3. Central nervous system tumor, metastasis(es), and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period or identified prior to consent.
4. Active infection requiring treatment.
5. Out-of-range laboratory values defined as:

   * Absolute neutrophil count (ANC) <1.5 × 10^9/L
   * Hemoglobin <9 g/dL
   * Platelets <100 × 10^9/L)
   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) >2.5 × the upper limit of normal (ULN) or ≥5 × ULN with liver involvement
   * Total bilirubin >1.5 × ULN
   * Serum creatinine >1.5 × ULN or creatinine clearance (CrCl≤60mL/min, measured or calculated using the Cockcroft-Gault Method
   * International Normalized Ratio (INR) or prothrombin time (PT) >1.5 × ULN and activated partial thromboplastin time (aPTT) >1.5 × ULN (unless patient is receiving anticoagulant therapy)
6. Inability to swallow oral medications or presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of MTB-9655 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, malabsorption syndrome).
7. Any of the following cardiac criteria:

   * Known history of marked prolongation of QT/corrected QT(QT/QTc) interval.
   * Clinically significant cardiovascular disease, including cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure,or serious uncontrolled cardiac arrhythmia requiring medication.
   * History of additional risk factors for Torsade de Pointes (including heart failure, hypokalemia, family history of long QT syndrome, and use of concomitant medications that prolong the QT/QTc interval.
   * Patients with a left ventricular ejection fraction (LVEF) <50%.
8. History of concomitant malignancy with recurrence <3 year from enrolment.
9. Expected to require any other form of systemic or localized antineoplastic therapy while on trial.
10. Significant liver cirrhosis defined as Child-Pugh Class B or C.
11. History of hemolytic disorders.
12. Active infection with human immunodeficiency virus (HIV).
13. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
14. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of participants with dose limiting toxicities (DLTs) from MTB-9655 monotherapy in patients with locally advanced or metastatic solid tumors. | 21 days
  DLTs are defined as adverse events (graded according to NCI CTCAE v5.0) during first 21 days of treatment that are related to MTB-9655 monotherapy
Part A: Maximum tolerated dose (MTD) by the number of participants with dose limiting toxicities (DLTs) from MTB-9655 monotherapy | At the end of Cycle 1 (each cycle is 21 days)
Recommended Phase 2 dose (RP2D) of MTB-9655 monotherapy in patients with locally advanced or metastatic solid tumors. | From Cycle 1 Day 1 until up to 30 days post last dose (each cycle is 21 days)
  The RP2D level will be no higher than the identified Maximum Tolerated Dose (MTD)
Number of participants with adverse events following administration of MTB-9655 | From Cycle 1 Day 1 until up to 30 days post last dose (each cycle is 21 days)
  Adverse events are graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetic Analysis single dose : maximum plasma concentration (Cmax) for MTB-9655 | 22 days ,from Cycle 0 to Cycle 2 Day1. Each cycle is 21 days.
  Blood samples will be collected for calculation of pharmacokinetic (PK) parameters.
Pharmacokinetic Analysis (multiple dose): Time to maximum plasma concentration at steady state (tmax ss) for MTB-9655 | 22 days -from Cycle 0 to Cycle 2 Day1. Each cycle is 21 days.
  Blood samples analyzed by biochemical assays at initial dose drug levels and steady -state drug levels.
Overall response rate in participants receiving MTB-9655 | Every 6 weeks from Cycle 1 Day1 for 24 weeks, then every 12 weeks up to 24 months (each cycle is 21 days)
  Overall response rate is defined as the proportion of patients who have a best response of either complete response (CR) or partial response (PR) based on RECIST v1.1
Duration of response based on RECIST 1.1 | Every 6 weeks from Cycle 1 Day 1 for 24 weeks, then every 12 weeks until disease progression or death or up to 1 year
  Duration of response will be defined for patients with a Best Overall Response of CR/PR as the time from the date of first documented response until date of documented progression (by RECIST v1.1), or death in the absence of disease progression.
Disease control rate based on RECIST 1.1 | Every 6 weeks from Cycle 1 Day 1 for 24 weeks, then every 12 weeks until disease progression or death or up to 1 year
  Disease control rate is defined as the proportion of patients with CR, PR, or SD based on RECIST v1.1
Progression free survival based on RECIST 1.1 | Every 6 weeks from Cycle 1 Day 1 for 24 weeks, then every 12 weeks until disease progression or death or up to 1 year
  Progression free survival is defined as the time from the start of study treatment until the earliest objective disease progression defined( by RECIST v1.1),or death by any cause in the absence of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith McKean, MD, Study Chair — SCRI Development Innovations, LLC
Locations (3):
- Tennessee Oncology, Nashville, Tennessee, United States
- Israel (2):
  - Rambam MC, Haifa
  - Sourasky MC, Tel Aviv

IPD SHARING:
Plan to Share IPD: No